CLINICAL TRIAL: NCT06668285
Title: The Effect of Parental Presence on the Child's Comfort and Physiologic Parameters in PICU
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, ESRA ARDAHAN AKGUL, Asst. Prof., Izmir Katip Celebi University
Other Study IDs: 101
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Family Centered Care; Comfort; Vital Sign Evaluation; Parent
Keywords: family centered care; parents presence; comfort; vital signs

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: parental presence — parental presence in PICU

SUMMARY:
The study was planned to be conducted and completed within 6 months after ethics committee approval was obtained. The research is a prospective, quasi-experimental study.

The population of the study will consist of children hospitalized in the Pediatric Intensive Care Unit of SBU, Izmir Dr. Behçet Uz Pediatric Diseases and Surgery Training and Research Hospital. Randomization of children will be done to determine which children's data will be followed on the relevant visit day.

Physiologic parameters including respiratory rate, pulse rate, oxygen saturation, body temperature, blood pressure and comfort levels of the children will be evaluated just before, during and after the parental visit (1st minute and 5th minute) and compared with those before the parental visit. All observations will be made by the same nurse to avoid bias in the study.

DETAILED DESCRIPTION:
There is a growing concern about psychological sequelae in children after hospitalization in the PICU. Despite the prevalence of adverse outcomes such as post-traumatic stress disorder, anxiety and behavioral problems in children after NICU admission, interventions to promote children's comfort have been limited. Children are physically and emotionally vulnerable and exposed to highly harmful environmental stimuli in the PICU. In a study by Johnston et al. in which mothers attempted to touch and talk to children during invasive procedures to reduce children's pain, children recovered faster and mothers experienced reduced anxiety, helplessness and an increased sense of purpose in caring for their children. Melnyk et al. examined the effect of a maternal coping intervention and found less anxiety in mothers and children. Despite these findings, the role of the parent when a child is hospitalized in the PICU is poorly defined. Parents describe the role change in the PICU as a tremendous stressor and report feeling helpless, anxious and fearful at the bedside. They suggest that comforting approaches that mimic home routines may alleviate these feelings and benefit their child.The study is planned to be conducted and completed within 6 months after ethics committee approval was obtained. The research is a prospective, quasi-experimental study.

The population of the study will consist of children hospitalized in the Pediatric Intensive Care Unit of SBU, Izmir Dr. Behçet Uz Pediatric Diseases and Surgery Training and Research Hospital. Randomization of children will be done to determine which children's data will be followed on the relevant visit day.

Physiologic parameters including respiratory rate, pulse rate, oxygen saturation, body temperature, blood pressure and comfort levels of the children will be evaluated just before, during and after the parental visit (1st minute and 5th minute) and compared with those before the parental visit. All observations will be made by the same nurse to avoid bias in the study

ELIGIBILITY:
Inclusion Criteria

1. Being hospitalized in Behçet Uz Pediatric Intensive Care Unit
2. Parent's volunteering to participate in the study Exclusion Criteria

1. Any intervention by the child's parent that may affect the dependent variables (watching cartoons, listening to music, etc.)

Ages: 0 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 0-3 years
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
comfort scale point | Baseline, and first minute of the visit and first/fifth minute after the visit
  before, during and after the 1st and 5th minute of the visit

SECONDARY OUTCOMES:
heart rate | Baseline, and first minute of the visit and first/fifth minute after the visit
  heart rate will be measured by Braun YK-81CEU
saturation | Baseline, and first minute of the visit and first/fifth minute after the visit
  saturation will be measured by Braun YK-81CEU
respiratory rate | Baseline, and first minute of the visit and first/fifth minute after the visit
  respiratory rate will be measured by Braun YK-81CEU
blood pressure | Baseline, and first minute of the visit and first/fifth minute after the visit
  blood pressure will be measured by Nimo HS-20C Aneroid

CONTACTS AND LOCATIONS:
Overall Officials: Esra Ardahan Akgül, PhD, Study Chair — İzmir Katip Çelebi University

IPD SHARING:
Plan to Share IPD: No